CLINICAL TRIAL: NCT06334068
Title: Short-term Glycemic Control in Patients With Uncontrolled Diabetes Mellitus Before Major Abdominal Surgery for Reducing Morbidity and Mortality: A Randomized Controlled Trial
Brief Title: SHOrt-term Glycemic Control for Reducing Post-SURGical Complications
Acronym: ShoGR-Surg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MS.24.03.2725
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Diabetes; Uncontrolled Diabtetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The patients in the preoperative anesthesia clinic are divided into one of the following groups:
  1. Short-term glycemic control group:
     Patients will be admitted to the hospital for 2-3 days before surgery. During this pilot study, patients will be admitted to the intermediate care unit to monitor and control preoperative blood glucose. We aim to maintain moderate glucose control (140 - 180 mg/dl) using basal-bolus insulin protocol plus correctional doses as needed.
  2. Standard-of-care group: Patients will be admitted the day before surgery with the usual patient treatment.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors, who will call patients or relatives 30 days after surgery, will be masked for the allocated group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short-term glycemic control group (Experimental): Patients will be admitted to the hospital for 2-3 days before surgery. During this pilot study, patients will be admitted to the intermediate care unit to monitor and control preoperative blood glucose. We aim to maintain moderate glucose control (140-180 mg/dl) using the basal-bolus insulin protocol, plus correctional doses as needed.
  Interventions: Other: Short-term glycemic control group
- Standard-of-care group (Active Comparator): Patients will be admitted the day before surgery with the usual patient treatment.
  Interventions: Other: Standard-of-care group

INTERVENTIONS:
Other: Short-term glycemic control group — Patients will be admitted to the hospital for 2-3 days before surgery. During this pilot study, patients will be admitted to the intermediate care unit to monitor and control preoperative blood glucose. We aim to maintain moderate glucose control (140-180 mg/dl) using the basal-bolus insulin protocol, plus correctional doses as needed.
  Other Names: Active Intervention
  Arms: Short-term glycemic control group
Other: Standard-of-care group — Patients will be admitted the day before surgery with the usual patient treatment.
  Other Names: Control group
  Arms: Standard-of-care group

SUMMARY:
Perioperative dysglycemia-hyperglycemia, hypoglycemia, and glycemic variability-is associated with an increased risk for adverse outcomes. Several studies have reported the association between elevated preoperative HbA1c and postoperative complications.

There are no studies that confirm that postponing elective surgery improves patient outcomes. Likewise, no prospective trials have studied whether short-term glycemic control reduces postoperative complications and unnecessary patient delays in elective surgeries.

Consequently, this randomized controlled trial aimed to investigate the effects of short-term glycemic control before major abdominal surgery on postoperative morbidity and mortality.

DETAILED DESCRIPTION:
Despite the limitations of measurements of HbA1c, guidelines for perioperative glycemic management suggest delaying elective surgery if HbA1c exceeds certain levels (7-8.5%) (Joshi et al., 2010; CPOC, 2022). However, no studies confirm that postponing elective surgery improves patient outcomes. Likewise, no prospective trials have studied whether short-term glycemic control reduces postoperative complications and unnecessary patient delays in elective surgeries (Duggan et al., 2017).

Consequently, this randomized controlled trial aimed to investigate the effects of short-term glycemic control before major abdominal surgery on postoperative morbidity and mortality. The study hypothesis is that in diabetic patients who are presenting for non-cardiac non-elective surgery and whose HbA1c is ≥7.5% (≥58 mmol/mol), short-term glycemic control would improve outcome compared to standard-of-care, as measured with days-at-home at 30 postoperative days (DAH-30).

The current study aims to detect the value of short-term glycemic control in uncontrolled diabetic patients (preoperative HbA1c ≥7.5% [≥58 mmol/mol]) for reducing postoperative morbidity and mortality.

The patients in the preoperative anesthesia clinic will be randomized into one of the upcoming groups:

1. Short-term glycemic control group:

   Patients will be admitted to the hospital for 2-3 days before surgery. During this pilot study, patients will be admitted to the intermediate care unit to monitor and control preoperative blood glucose. We aim to maintain moderate glucose control (140 - 180 mg/dl) using basal-bolus insulin protocol plus correctional doses as needed.
2. Standard-of-care group: Patients will be admitted the day before surgery with the usual patient treatment.

In both groups, diabetic drugs will be managed per local protocol.

ELIGIBILITY:
Inclusion Criteria:

* all adult diabetic patients (≥18 years) of either sex scheduled for major abdominal surgery (estimated operative time is > 2 hours) with Hb A1c ≥7.5% (58 mmol/mol).

Exclusion Criteria:

* Patients < 18 years
* Emergency Surgery
* Elective surgery that can be postponed safely till glycemic control
* Hb A1c < 7.5%
* Pregnant patients
* Patient Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-02-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Number of days at home after surgery (DAH-30). | 30 days after surgery
  Continuous outcome as the number of days over the 30 days after surgery.

SECONDARY OUTCOMES:
Loss of follow-up after surgery | 30 days after Surgery
  Incidence (yes/no) outcome
Loss of follow up after the clinic preoperative assessment | 30 days after initial assessment
  incidence (yes/no) outcome
30-day mortality | 30 days after surgery
  incidence (yes/no) outcome
Length of hospital stay | 30 days after surgery
  continuous outcome: number of days untill discharge from hospital after surgery
incidence of postoperative complications | 30 days after surgery
  according to the comprehensive complications index (Kalt et al., 2023)
Quality of Recovery15 (QoR-15) | after 24 hours of surgery
  a score of 15 items
clinic-to-admission and clinic-to-surgery intervals | 30 days
  The time interval between the preoperative anesthesia clinic and admission or surgery in days, respectively.

OTHER OUTCOMES:
Time to resumption of normal diabetes therapy | 60 days after surgery
  number in days
Incidence of diabetic ketoacidosis or hypoglycemia | during the hospitalization period (within 30 days after surgery)
  incidence (yes/no) outcome
Incidence of use of intravenous insulin infusion therapy | during the hospitalization period (within 30 days after surgery)
  incidence (yes/no) outcome
Duration of use of intravenous insulin infusion therapy | during the hospitalization period (within 30 days after surgery)
  duration in days and hours
Change in diabetic management at 30 days | during the hospitalization period (after 30 days after surgery)
  incidence (yes/no) outcome

CONTACTS AND LOCATIONS:
Overall Officials: Moataz M Emara, MD, EDAIC, Principal Investigator — Mansoura University Hospital
Locations (1):
- Moataz Maher Emara, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The anonymized individual data will be available with the principal investigator on reasonable request after IRB approval within two years of publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Will be reported as soon as possible.
Access Criteria: Will be reported as soon as possible.